CLINICAL TRIAL: NCT02217878
Title: A Randomized, Double-blind Study Evaluating the Influence of Morphine on Pharmacokinetics and Pharmacodynamics of Ticagrelor and Its Active Metabolite (AR-C124910XX) in Patients With ST-segment Elevation Myocardial Infarction and Non-ST-segment Elevation Myocardial Infarction.
Brief Title: Influence of Morphine on Pharmacokinetics and Pharmacodynamics of Ticagrelor in Patients With Acute Myocardial Infarction
Acronym: IMPRESSION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Prof. dr hab., Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUMK202
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: ST-segment Elevation Myocardial Infarction; Non-ST-segment Elevation Myocardial Infarction; VA Drug Interactions
Keywords: ST-segment elevation myocardial infarction; non-ST-segment elevation myocardial infarction; ticagrelor; morphine; pharmacokinetics; pharmacodynamics; drug interactions; VASP assay; Multiple Electrode Aggregometry; VerifyNow
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Morphine; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Active Comparator): morphine sulfate 5 mg IV followed by 180 mg loading dose of ticagrelor
  Interventions: Drug: Morphine; Drug: Ticagrelor
- Placebo (Placebo Comparator): sodium chloride 0,9% 5 mg IV followed by 180 mg loading dose of ticagrelor
  Interventions: Drug: Placebo; Drug: Ticagrelor

INTERVENTIONS:
Drug: Morphine — IV bolus injection
  Other Names: Morphine sulfate
  Arms: Morphine
Drug: Placebo — IV bolus injection
  Other Names: Sodium chloride 0,9%
  Arms: Placebo
Drug: Ticagrelor — 180 mg loading dose
  Other Names: Brilique

SUMMARY:
The purpose of the IMPRESSION study is to determine whether intravenous administration of morphine prior to ticagrelor administration in ST-segment elevation myocardial infarction (STEMI) patients and in non-ST-segment elevation myocardial infarction (NSTEMI) patients alters the plasma concentrations of ticagrelor and its active metabolite and whether it is associated with any negative impact on the antiplatelet effect of ticagrelor.

DETAILED DESCRIPTION:
The European Society of Cardiology and American Heart Association guidelines recommend use of morphine as a treatment of choice for pain relief in STEMI patients. However, this recommendation, although strong, is only based on expert consensus (class of recommendation I, level of evidence C). Morphine, apart from its analgesic effects, also alleviates the work of breathing and reduces anxiety. On the other hand, despite its favorable analgesic and sedative actions, morphine also exerts adverse effects, which include hypotension, bradycardia, respiratory depression, vomiting and reduction of gastrointestinal motility. Some of the previously listed morphine's side effects could affect the intestinal absorption and thus pharmacokinetics and pharmacodynamics of orally administered drugs which are concomitantly used with morphine. At present, no pharmacokinetic and pharmacodynamic data regarding the concurrent use of morphine and P2Y12 blockers in the STEMI or NSTEMI setting are available. Therefore, evidence-based verification of morphine's influence on pharmacokinetics and pharmacodynamics of ticagrelor and its active metabolite (AR-C124910XX) could provide a valuable insight in the knowledge regarding modern acute myocardial infarction management.

Predefined subanalysis: aimed to investigate which one of platelet reactivity assessment methods utilized in the study (VASP assay, MEA, LTA, VerifyNow) best reflects concentration of ticagrelor and its active metabolite (AR-C124910XX).

Since there is no reference study examining pharmacokinetics of ticagrelor in STEMI or NSTEMI patients, we decided to perform an internal pilot study of approximately 30 patients (15 patients for each arm) for estimating the final sample size.

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent prior to any study specific procedures
* diagnosis of acute ST-segment elevation myocardial infarction or acute non-ST-segment elevation myocardial infarction
* male or non-pregnant female, aged 18-80 years old
* provision of informed consent for angiography and PCI

Exclusion Criteria:

* chest pain described by the patient as unbearable or patient's request for analgesics
* prior morphine administration during the current STEMI or NSTEMI
* treatment with ticlopidine, clopidogrel, prasugrel or ticagrelor within 14 days before the study enrollment
* hypersensitivity to ticagrelor
* current treatment with oral anticoagulant or chronic therapy with low-molecular-weight heparin
* active bleeding
* history of intracranial hemorrhage
* recent gastrointestinal bleeding (within 30 days)
* history of coagulation disorders
* platelet count less than <100 x10^3/mcl
* hemoglobin concentration less than 10.0 g/dl
* history of moderate or severe hepatic impairment
* history of major surgery or severe trauma (within 3 months)
* patients considered by the investigator to be at risk of bradycardic events
* second or third degree atrioventricular block during screening for eligibility
* history of asthma or severe chronic obstructive pulmonary disease
* patient required dialysis
* manifest infection or inflammatory state
* Killip class III or IV during screening for eligibility
* respiratory failure
* history of severe chronic heart failure (NYHA class III or IV)
* concomitant therapy with strong CYP3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir) or strong CYP3A inducers (rifampicin, phenytoin, carbamazepine, dexamethasone, phenobarbital) within 14 days and during study treatment
* body weight below 50 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Jacek Kubica, MD, PhD, Principal Investigator — Collegium Medicum im. Ludwika Rydygiera w Bydgoszczy, Uniwersytet Mikołaja Kopernika w Toruniu
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kubica J, Adamski P, Ostrowska M, Sikora J, Kubica JM, Sroka WD, Stankowska K, Buszko K, Navarese EP, Jilma B, Siller-Matula JM, Marszall MP, Rosc D, Kozinski M. Morphine delays and attenuates ticagrelor exposure and action in patients with myocardial infarction: the randomized, double-blind, placebo-controlled IMPRESSION trial. Eur Heart J. 2016 Jan 14;37(3):245-52. doi: 10.1093/eurheartj/ehv547. Epub 2015 Oct 21. PMID 26491112
- [Derived] Kubica J, Adamski P, Ostrowska M, Kozinski M, Obonska K, Laskowska E, Obonska E, Grzesk G, Winiarski P, Paciorek P. Influence of Morphine on Pharmacokinetics and Pharmacodynamics of Ticagrelor in Patients with Acute Myocardial Infarction (IMPRESSION): study protocol for a randomized controlled trial. Trials. 2015 Apr 29;16:198. doi: 10.1186/s13063-015-0724-z. PMID 25925591

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morphine | Placebo
Started | 37 | 37
Completed | 35 | 35
Not Completed | 2 | 2
Not completed — required morphine due to chest pain | 1 | 2
Not completed — initial diagnosis of STEMI not confirmed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.5) | 62.5 (10.5) | 61.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 23 | 28 | 51
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (4.3) | 27.4 (4.0) | 27.5 (4.2)
STEMI [Number; unit: participants] | 24 | 21 | 45
GP IIb/IIIa administration [Number; unit: participants] | 10 | 6 | 16
Hypertension [Number; unit: participants] | 15 | 21 | 36
Diabetes mellitus [Number; unit: participants] | 8 | 5 | 13
Dyslipidaemia [Number; unit: participants] | 30 | 31 | 61
Current smoker [Number; unit: participants] | 17 | 14 | 31
Prior AMI [Number; unit: participants] | 5 | 8 | 13
Prior PCI [Number; unit: participants] | 4 | 9 | 13
Prior CABG [Number; unit: participants] | 0 | 0 | 0
Prior non-severe heart failure [Number; unit: participants] | 0 | 3 | 3
Prior non-haemorrhagic stroke [Number; unit: participants] | 1 | 0 | 1
Peripheral arterial disease [Number; unit: participants] | 3 | 1 | 4
Chronic renal disease [Number; unit: participants] | 1 | 2 | 3
Chronic obstructive pulmonary disease [Number; unit: participants] | 2 | 0 | 2
Gout [Number; unit: participants] | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve for Ticagrelor (AUC 0-12h)
Description: Exposure to ticagrelor during the first 12 hours after ticagrelor loading dose
Time Frame: prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h, 12h post dose
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
ng*h/mL | 6307 (4359) | 9791 (5136)

2. Secondary Outcome: Area Under the Plasma Concentration-time Curve for AR-C124910XX (AUC 0-12h)
Description: Exposure to ticagrelor metabolite during the first 12 hours after ticagrelor loading dose
Time Frame: prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h, 12h post dose
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
ng*h/mL | 1503 (1138) | 2388 (1555)

3. Secondary Outcome: Maximum Concentration of Ticagrelor
Description: Maximum concentration (Cmax) of ticagrelor
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
ng/mL | 1156 (771) | 1683 (847)

4. Secondary Outcome: Maximum Concentration of AR-C124910XX
Description: Maximum concentration (Cmax) of AR-C124910XX
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
ng/mL | 1085 [508 to 1709] | 1043 [792 to 1572]

5. Secondary Outcome: Time to Maximum Concentration for Ticagrelor
Description: Time to maximum concentration (Tmax) for ticagrelor
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
hours | 4 [3 to 12] | 2 [2 to 4]

6. Secondary Outcome: Time to Maximum Concentration for AR-C124910XX
Description: Time to maximum concentration (Tmax) for AR-C124910XX
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
hours | 4 [3 to 12] | 4 [3 to 6]

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve for Ticagrelor (AUC 0-6h)
Description: Exposure to ticagrelor during the first 6 hours after ticagrelor loading dose
Time Frame: prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h post dose
Measure: Median (Inter-Quartile Range); unit: ng*h/mL
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
ng*h/mL | 2491 [189 to 5764] | 5587 [2810 to 8546]

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve for AR-C124910XX (AUC 0-6)
Description: Exposure to ticagrelor metabolite during the first 6 hours after ticagrelor loading dose
Time Frame: prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h post dose
Measure: Median (Inter-Quartile Range); unit: ng*h/mL
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
ng*h/mL | 472 [0 to 1036] | 1001 [643 to 1666]

9. Secondary Outcome: Platelet Reactivity Index Assessed by VASP Assay
Description: Platelet Reactivity Index (PRI) evaluated by VASP assay (cut-off value for high platelet reactivity: PRI >50%)
Time Frame: prior to the initial ticagrelor dose
Measure: Median (Inter-Quartile Range); unit: Platelet Reactivity Index (%)
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
Platelet Reactivity Index (%) | 88.5 [82.9 to 93.5] | 88.3 [81.5 to 94.0]

10. Secondary Outcome: Platelet Reactivity Index Assessed by VASP Assay
Description: Platelet Reactivity Index (PRI) evaluated by VASP assay (cut-off value for high platelet reactivity: PRI >50%)
Time Frame: 30 minutes post ticagrelor dose
Measure: Median (Inter-Quartile Range); unit: Platelet Reactivity Index (%)
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
Platelet Reactivity Index (%) | 83.2 [74.5 to 89.7] | 73.9 [42.6 to 87.7]

11. Secondary Outcome: Platelet Reactivity Index Assessed by VASP Assay
Description: Platelet Reactivity Index (PRI) evaluated by VASP assay (cut-off value for high platelet reactivity: PRI >50%)
Time Frame: 1 hour post ticagrelor dose
Measure: Median (Inter-Quartile Range); unit: Platelet Reactivity Index (%)
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
Platelet Reactivity Index (%) | 70.2 [34.1 to 87.2] | 42.0 [25.6 to 81.2]

12. Secondary Outcome: Platelet Reactivity Index Assessed by VASP Assay
Description: Platelet Reactivity Index (PRI) evaluated by VASP assay (cut-off value for high platelet reactivity: PRI >50%)
Time Frame: 2 hours post ticagrelor dose
Measure: Median (Inter-Quartile Range); unit: Platelet Reactivity Index (%)
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
Platelet Reactivity Index (%) | 52.1 [21.7 to 80.5] | 26.2 [18.7 to 52.1]

13. Secondary Outcome: Platelet Reactivity Index Assessed by VASP Assay
Description: Platelet Reactivity Index (PRI) evaluated by VASP assay (cut-off value for high platelet reactivity: PRI >50%)
Time Frame: 3 hours post ticagrelor dose
Measure: Median (Inter-Quartile Range); unit: Platelet Reactivity Index (%)
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
Platelet Reactivity Index (%) | 37.8 [24.7 to 75.1] | 26.0 [13.1 to 52.4]

14. Secondary Outcome: Platelet Reactivity Index Assessed by VASP Assay
Description: Platelet Reactivity Index (PRI) evaluated by VASP assay (cut-off value for high platelet reactivity: PRI >50%)
Time Frame: 4 hours post ticagrelor dose
Measure: Median (Inter-Quartile Range); unit: Platelet Reactivity Index (%)
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
Platelet Reactivity Index (%) | 36.9 [19.1 to 64.1] | 23.2 [14.3 to 43.4]

15. Secondary Outcome: Platelet Reactivity Index Assessed by VASP Assay
Description: Platelet Reactivity Index (PRI) evaluated by VASP assay (cut-off value for high platelet reactivity: PRI >50%)
Time Frame: 6 hours post ticagrelor dose
Measure: Median (Inter-Quartile Range); unit: Platelet Reactivity Index (%)
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
Platelet Reactivity Index (%) | 27.9 [18.2 to 44.1] | 19.7 [12.7 to 33.0]

16. Secondary Outcome: Platelet Reactivity Index Assessed by VASP Assay
Description: Platelet Reactivity Index (PRI) evaluated by VASP assay (cut-off value for high platelet reactivity: PRI >50%)
Time Frame: 12 hours post ticagrelor dose
Measure: Median (Inter-Quartile Range); unit: Platelet Reactivity Index (%)
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
Platelet Reactivity Index (%) | 27.5 [17.0 to 42.3] | 15.6 [12.3 to 33.1]

17. Secondary Outcome: Platelet Arbitrary Aggregation Units Assessed by Multiple Electrode Aggregometry
Description: Platelet reactivity assessed by Multiple Electrode Aggregometry (cut-off value for high platelet reactivity: AUC >46 Platelet Arbitrary Aggregation Units)
Time Frame: prior to the initial ticagrelor dose
Population: According to the study protocol multiple electrode aggregometry pharmacodynamic evaluation was performed in all patients except for those treated with glycoprotein (GP) IIb/IIIa receptor inhibitors.
Measure: Median (Inter-Quartile Range); unit: Platelet Arbitrary Aggregation Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 29
Platelet Arbitrary Aggregation Units | 85 [70 to 102] | 77 [54 to 95]

18. Secondary Outcome: Platelet Arbitrary Aggregation Units Assessed by Multiple Electrode Aggregometry
Description: as for outcome 17
Time Frame: 30 minutes post ticagrelor dose
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Platelet Arbitrary Aggregation Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 29
Platelet Arbitrary Aggregation Units | 86 [53 to 99] | 48 [22 to 89]

19. Secondary Outcome: Platelet Arbitrary Aggregation Units Assessed by Multiple Electrode Aggregometry
Description: as for outcome 17
Time Frame: 1 hour post ticagrelor dose
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Platelet Arbitrary Aggregation Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 29
Platelet Arbitrary Aggregation Units | 59 [31 to 86] | 23 [17 to 60]

20. Secondary Outcome: Platelet Arbitrary Aggregation Units Assessed by Multiple Electrode Aggregometry
Description: as for outcome 17
Time Frame: 2 hours post ticagrelor dose
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Platelet Arbitrary Aggregation Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 29
Platelet Arbitrary Aggregation Units | 31 [20 to 71] | 23 [10 to 36]

21. Secondary Outcome: Platelet Arbitrary Aggregation Units Assessed by Multiple Electrode Aggregometry
Description: as for outcome 17
Time Frame: 3 hours post ticagrelor dose
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Platelet Arbitrary Aggregation Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 35
Platelet Arbitrary Aggregation Units | 27 [18 to 55] | 17 [10 to 23]

22. Secondary Outcome: Platelet Arbitrary Aggregation Units Assessed by Multiple Electrode Aggregometry
Description: as for outcome 17
Time Frame: 4 hours post ticagrelor dose
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Platelet Arbitrary Aggregation Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 29
Platelet Arbitrary Aggregation Units | 29 [10 to 44] | 13 [9 to 22]

23. Secondary Outcome: Platelet Arbitrary Aggregation Units Assessed by Multiple Electrode Aggregometry
Description: as for outcome 17
Time Frame: 6 hours post ticagrelor dose
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Platelet Arbitrary Aggregation Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 29
Platelet Arbitrary Aggregation Units | 19 [9 to 34] | 11 [5 to 15]

24. Secondary Outcome: Platelet Arbitrary Aggregation Units Assessed by Multiple Electrode Aggregometry
Description: as for outcome 17
Time Frame: 12 hours post ticagrelor dose
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Platelet Arbitrary Aggregation Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 29
Platelet Arbitrary Aggregation Units | 19 [10 to 27] | 11 [7 to 16]

25. Secondary Outcome: P2Y12 Reaction Units Assessed by VerifyNow
Description: P2Y12 Reaction Units (PRU) Assessed by VerifyNow (cut-off value for high platelet reactivity: PRU >208)
Time Frame: prior to the initial ticagrelor dose
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Median (Inter-Quartile Range); unit: P2Y12 Reaction Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
P2Y12 Reaction Units | 232.5 [197.0 to 270.0] | 238.5 [194.0 to 267.0]

26. Secondary Outcome: P2Y12 Reaction Units Assessed by VerifyNow
Description: P2Y12 Reaction Units (PRU) Assessed by VerifyNow (cut-off value for high platelet reactivity: PRU >208)
Time Frame: 30 minutes post ticagrelor dose
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Median (Inter-Quartile Range); unit: P2Y12 Reaction Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
P2Y12 Reaction Units | 268.5 [202.0 to 299.0] | 210.5 [118.0 to 266.0]

27. Secondary Outcome: P2Y12 Reaction Units Assessed by VerifyNow
Description: P2Y12 Reaction Units (PRU) Assessed by VerifyNow (cut-off value for high platelet reactivity: PRU >208)
Time Frame: 1 hour post ticagrelor dose
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Median (Inter-Quartile Range); unit: P2Y12 Reaction Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
P2Y12 Reaction Units | 206.5 [88.0 to 266.0] | 117.0 [10.0 to 233.0]

28. Secondary Outcome: P2Y12 Reaction Units Assessed by VerifyNow
Description: P2Y12 Reaction Units (PRU) Assessed by VerifyNow (cut-off value for high platelet reactivity: PRU >208)
Time Frame: 2 hours post ticagrelor dose
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Median (Inter-Quartile Range); unit: P2Y12 Reaction Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
P2Y12 Reaction Units | 137.0 [27.0 to 251.0] | 44.0 [7.0 to 119.0]

29. Secondary Outcome: P2Y12 Reaction Units Assessed by VerifyNow
Description: P2Y12 Reaction Units (PRU) Assessed by VerifyNow (cut-off value for high platelet reactivity: PRU >208)
Time Frame: 3 hours post ticagrelor dose
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Median (Inter-Quartile Range); unit: P2Y12 Reaction Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
P2Y12 Reaction Units | 113.0 [31.0 to 221.0] | 15.0 [4.0 to 52.0]

30. Secondary Outcome: P2Y12 Reaction Units Assessed by VerifyNow
Description: P2Y12 Reaction Units (PRU) Assessed by VerifyNow (cut-off value for high platelet reactivity: PRU >208)
Time Frame: 4 hours post ticagrelor dose
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Median (Inter-Quartile Range); unit: P2Y12 Reaction Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
P2Y12 Reaction Units | 50.5 [8.0 to 165.0] | 9.0 [4.0 to 72.0]

31. Secondary Outcome: P2Y12 Reaction Units Assessed by VerifyNow
Description: P2Y12 Reaction Units (PRU) Assessed by VerifyNow (cut-off value for high platelet reactivity: PRU >208)
Time Frame: 6 hours post ticagrelor dose
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Median (Inter-Quartile Range); unit: P2Y12 Reaction Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
P2Y12 Reaction Units | 44.5 [6.0 to 171.0] | 8.0 [3.0 to 21.0]

32. Secondary Outcome: P2Y12 Reaction Units Assessed by VerifyNow
Description: P2Y12 Reaction Units (PRU) Assessed by VerifyNow (cut-off value for high platelet reactivity: PRU >208)
Time Frame: 12 hours post ticagrelor dose
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Median (Inter-Quartile Range); unit: P2Y12 Reaction Units
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
P2Y12 Reaction Units | 9.0 [4.0 to 116.0] | 7.5 [3.0 to 48.0]

33. Secondary Outcome: Percentage of Patients With High Platelet Reactivity After the Loading Dose of Ticagrelor Assessed With VASP
Description: Percentage of Patients With High Platelet Reactivity (HPR) After the Loading Dose of Ticagrelor Assessed With VASP
Time Frame: 2 hours
Measure: Number; unit: Percentage of Patients With HPR
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
Percentage of Patients With HPR | 57 | 29

34. Secondary Outcome: Percentage of Patients With High Platelet Reactivity After the Loading Dose of Ticagrelor Assessed With MEA
Description: Percentage of Patients With High Platelet Reactivity (HPR) After the Loading Dose of Ticagrelor Assessed With MEA
Time Frame: 2 hours
Population: as for outcome 17
Measure: Number; unit: Percentage of Patients With HPR
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 29
Percentage of Patients With HPR | 40 | 14

35. Secondary Outcome: Percentage of Patients With High Platelet Reactivity After the Loading Dose of Ticagrelor Assessed With VerifyNow
Description: Percentage of Patients With High Platelet Reactivity (HPR) After the Loading Dose of Ticagrelor Assessed With VerifyNow
Time Frame: 2 hours
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Number; unit: Percentage of Patients With HPR
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
Percentage of Patients With HPR | 36 | 19

36. Secondary Outcome: Time to Reach Platelet Reactivity Below the Cut-off Value for High Platelet Reactivity Evaluated With VASP
Description: Time to Reach Platelet Reactivity Below the Cut-off Value for High Platelet Reactivity (HPR) Evaluated With VASP
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 35 | 35
hours | 2.0 [1.0 to 6.0] | 1 [0.5 to 3]

37. Secondary Outcome: Time to Reach Platelet Reactivity Below the Cut-off Value for High Platelet Reactivity Evaluated With MEA
Description: Time to Reach Platelet Reactivity Below the Cut-off Value for High Platelet Reactivity (HPR) Evaluated With MEA
Time Frame: 12 hours
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 25 | 29
hours | 2.0 [1.0 to 4.0] | 1.0 [0.5 to 2.0]

38. Secondary Outcome: Time to Reach Platelet Reactivity Below the Cut-off Value for High Platelet Reactivity Evaluated With VerifyNow
Description: Time to Reach Platelet Reactivity Below the Cut-off Value for High Platelet Reactivity (HPR) Evaluated With VerifyNow
Time Frame: 12 hours
Population: In line with the study protocol, VerifyNow pharmacodynamic evaluation involved >30% of the overall study population.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 26 | 35
hours | 1.0 [0 to 3.0] | 0.5 [0 to 1.0]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Morphine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/35 | 2/35
Other Adverse Events (participants affected / at risk) | 5/35 | 7/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Morphine (N=35) | Placebo (N=35)
Stent thrombosis (Vascular disorders) | 1 | 0
Pulmonary oedema (Cardiac disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Morphine (N=35) | Placebo (N=35)
TIMI minor bleeding (Vascular disorders) | 0 | 4
TIMI minimal bleeding (Vascular disorders) | 0 | 1
Bradyarrhythmic event (Cardiac disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No